CLINICAL TRIAL: NCT07027384
Title: Evaluation of Digital Decision-support Tool for Child Nutritional Monitoring: a Protocol for Cluster Randomized Controlled Trial in Urban and Semi-Urban Areas in Indonesia
Acronym: KSI-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Indonesia's Strategic Development Initiatives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: koneksiRCT; 1447/CRG/2024/46-CISDI (Other Grant/Funding Number: KONEKSI)
Record Dates: First submitted 2025-06-09; First posted 2025-06-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Primary Health Care for Children; Nutritional Status
Keywords: mHealth; decision-support tools; community health workers; primary health care; posyandu

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web-Based App (Active Comparator): The first group of Posyandu will use the standard web-based version of the PN PRIMA app in addition to the routine nutritional services. This web-based version is accessible only through browsers and includes the basic functions such as reporting key health indicators and in-app warning alerts. This group will serve as the control group, using the baseline functionality of the app currently available to Kader
  Interventions: Device: Web-Based Apps PRIMA
- Mobile-Based App (Experimental): This group will receive access to the mobile version of PN PRIMA app. The mobile-based version has additional features unavailable in the web-based version. The mobile-based version has access to the PN PRIMA app using a standalone mobile app. In addition to the standard reporting of patients' key health indicators and in-app warning message alerts which are available in the web-based version, the mobile app includes active notifications for Kader, which serve as reminders to encourage Kader in making on-time assistance for healthcare beneficiaries, especially those considered requiring special attention (kunjungan khusus) and for those facing access barriers who need regular checkups (kunjungan rutin).
  Interventions: Device: Apps PRIMA Mobile
- Mobile + GEDSI Training (Experimental): In addition to using the new mobile-app as arm 2, this arm will include training module that focuses on identifying and addressing caregiver and community vulnerabilities. This training is designed to strengthen Kader's capacity in recognizing risk factors that may contribute to malnutrition, such as social, economic, and environmental barriers to care. The training emphasizes empathetic and responsive service delivery, equipping Kader not only with technological tools but also with improved understanding and skills for working in complex community settings. This integrated intervention enables the study to assess the combined effect of digital tools and conventional capacity-building efforts on service delivery outcomes.
  Interventions: Device: Apps PRIMA Mobile; Behavioral: Advance GEDSI Training

INTERVENTIONS:
Device: Web-Based Apps PRIMA — Apps PRIMA (posyandu monitoring tools) is delivered using a web-based app accessible through web browsers with basic core functionalities
  Arms: Web-Based App
Device: Apps PRIMA Mobile — Enhancement of Apps PRIMA delivered using a standalone mobile app. Enhanced core functionalities include the looping system of children measurements, automatic charts, and GEDSI-sensitive features
  Arms: Mobile + GEDSI Training; Mobile-Based App
Behavioral: Advance GEDSI Training — Additional training to address vulnerabilities in communities and empathetic service from CHWs to caregivers. The training is a follow-up training from a basic GEDSI materials already delivered to CHWs
  Arms: Mobile + GEDSI Training

SUMMARY:
This research is a collaborative study between Indonesia's Strategic Development Initiatives (CISDI), Knowledge Partnership Platform Australia - Indonesia (KONEKSI), Center on Child Protection and Wellbeing (PUSKAPA), and Center for Development Economics and Sustainability at Monash University. This study is a part of the PN PRIMA research universe, which is a program lead by CISDI with a focus of strengthening the primary healthcare facilities of Indonesia, known as Integrated Health Posts (Posyandu). This project supports the Ministry of Health's (MoH) flagship program: the Integrated Primary Health Care Services (ILP).

This study aims to evaluate the impact of implementing a digital mHealth app, called the PN PRIMA app, in enhancing the work quality of Community Health Workers working in Posyandu, known as Kader. This study specifically improve the PN PRIMA app from a web-based platform to a mobile application. We aim to improve data quality, streamline service delivery workflows, and enhance decision-making support for community health workers. The enhanced version incorporates new features and Gender Equality, Disability, and Social Inclusion (GEDSI) framework to strengthen primary health care delivery.

Impact evaluation of the study will be conducted through a three-arm parallel cluster randomized controlled trial. Posyandu will be the unit in which randomization will occur. The primary outcomes focuses on the improvements of Kader Posyandu performance in delivering follow-up home visits and how the app effectively support Kader in delivering nutrition interventions for children under five years of age.

The study will be conducted in the Puskesmas PN PRIMA catchment area, located in Kabupaten Bekasi and Kota Depok, focusing the intervention at the Posyandu level. In total, 38 Posyandu out of 12 health centers (Puskesmas) across the two areas will be recruited to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Community Health Workers (CHWs) assigned to work in one of the eligible Posyandu PN PRIMA
* Consent to participate in the program and the study

Exclusion Criteria:

- Community Health Workers working outside of Posyandu PN PRIMA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1030 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Completed follow-up home visits delivered as protocol | From intervention roll-out to the end of intervention period in 6 months
  Proportion of completed follow-up home visits that are delivered in a timely manner

SECONDARY OUTCOMES:
First follow-up home visitations | From intervention roll-out to the end of intervention period in 6 months
  Proportion of first follow-up visitations done within a week range following confirmation of cases from health workers
Knowledge and Attitude of CHWs | Measured in baseline (pre-intervention; maximum 1 months before training intervention) and endline (post-intervention; minimum 6 months intervention implementation)
  Kader's knowledge on children's nutritional needs and status, and attitudes toward vulnerable population
Caregiver's knowledge and attitude | Measured in baseline (pre-intervention; maximum 1 months before training intervention) and endline (post-intervention; minimum 6 months intervention implementation)
  Parents/caregivers knowledge on children's nutrition and primary care services, and attitudes towards primary healthcare services
Caregiver's satisfaction on healthcare | Measured in baseline (pre-intervention; maximum 1 months before training intervention) and endline (post-intervention; minimum 6 months intervention implementation)
  Parents/caregivers satisfaction towards primary healthcare services

OTHER OUTCOMES:
Feasibility on mHealth decision-support | Measured in endline (post-intervention) after 6 months
  Perception of feasibility and usability of apps PRIMA from Kader
Satisfaction on digital app | Measured in endline (post-intervention) after 6 months
  Satisfaction of digital app (apps PRIMA) by Kader

CONTACTS AND LOCATIONS:
Locations (6):
- Indonesia (6):
  - Puskesmas Sukmajaya, Depok, West Java
  - Puskesmas Abadijaya, Depok
  - Puskesmas Baktijaya, Depok
  - Puskesmas Cinangka, Depok
  - Puskesmas Limo, Depok
  - Puskesmas Sukatani, Depok